CLINICAL TRIAL: NCT05495035
Title: Study for Safety and Efficacy Evaluation of Olverembatinib Combined With APG-2575 in Children With Relapsed/Refractory Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia (R/R Ph + ALL）
Brief Title: Study for Safety and Efficacy of Olverembatinib Combined With APG-2575 in Children With Relapsed/Refractory Ph + ALL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HQP1351ACE01
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2022-08

CONDITIONS: Lymphoblastic Leukemia, Acute, Childhood; Leukemia, Lymphoblastic, Acute, Philadelphia-Positive; Relapsed Leukemia; Refractory Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — olverembatinib; Lisaftoclax; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olverembatinib + APG-2575 combinational therapy (Experimental): * Period 1: Olverembatinib alone period (2 weeks):
  * Period 2: olverembatinib in combination with APG-2575 and dexamethasone (4 weeks):
  Interventions: Drug: Olverembatinib, APG-2575, Dexamethasone

INTERVENTIONS:
Drug: Olverembatinib, APG-2575, Dexamethasone — * Period 1: Subjects will orally take olverembatinib 40mg adult equivalent dose alone QOD from Day 1 to Day 14 (D1 - D14) =. The investigator may start the combination therapy in advance based on medical conditions of the subjects, but not earlier than Day 5/the third dose (D5).
  * Period 2: 1) Subjects will orally take olverembatinib 40mg adult equivalent dose QOD from Day 15 to Day 42 (D15 - D42)).
    2) Subjects will orally take APG-2575 at a ramp up 200mg/400mg/600mg adult equivalent dos QD from D13 to D42 at a dose . In addition, a 3-day dose escalation from D13 to D15 will be needed, and the designated reference dose will be reached on D15.
    3) Subjects will orally take dexamethasone 6 mg/m2/day, QD from D15 to D42 at 6 mg/m2/day.

SUMMARY:
This is an open-label, multicenter, phase 1b study, which is designed to explore the safety, efficacy and PK of olverembatinib, a third-generation tyrosine kinase inhibitor (TKI) marketed in China, in combination with APG-2575 in treating R/R Ph+ALL children, and to preliminarily establish the recommended dose of olverembatinib and APG-2575 for children based on the above results.

DETAILED DESCRIPTION:
Eligible patients will receive a 6-week core treatment after screening, including a 2-week olverembatinib monotherapy and a 4-week combination therapy with olverembatinib, APG-2575 and dexamethasone, and based on the remission of leukemia after 2, 4, and 6 weeks of treatment, these patients will either continue olverembatinib alone/in combination with APG-2575 and dexamethasone as maintenance therapy or switch to other anti-tumor therapy.

Toxicities of this study will be graded according to NCI CTCAT (Version 5.0). The investigator will interrupt, reduce or discontinue the dose of the investigational drug according to the correlation and grade of toxicities. The study drug can be resumed when the drug related toxicities resolve to grade 1 or below.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients must meet all of the following criteria:

  1. Children under 18 years of age on the day of signing the informed consent form, and able to swallow the oral drugs during the study period.
  2. Subjects who are diagnosed with Ph+ALL, and are resistant or intolerant to at least one TKI. If the subject has BCR-ABL1 T315I mutation, prior use of TKIs will not be considered.

     Drug resistance includes disease recurrence and refractory disease. Relapse: Presence of blasts > 5% in peripheral blood or bone marrow or presence of extramedullary disease following CR. Refractory disease: Failure to have CR or incomplete remission (CRi) at the end of induction therapy. Intolerance refers to ≥ grade 3 non-hematological toxicity or ≥ grade 4 hematological toxicity in subjects which is at least possibly related to the last TKI treatment, lasts for > 2 weeks, and leads to TKI withdrawal.
  3. Informed consent of parents or legal guardians should be obtained before any study activities.
  4. For patients >16 years of age, Karnofsky performance status score ≥ 50; for patients ≤ 16 years of age, Lansky performance status score ≥ 50.
  5. Life expectancy of ≥ 3 months.
  6. For female patients of childbearing potential, urine β-HCG is negative.
  7. The following laboratory values must be met (reference ranges based on age and gender of children):

     1. Estimated glomerular filtration rate (eGFR) or radioisotope glomerular filtration rate (GFR) ≥70 mL/min/1.73 m2 based on Schwartz formula, or normal serum creatinine determined based on age and gender
     2. Serum albumin ≥ 3.0 g/dL
     3. Total bilirubin < 1.5 × upper limit of normal (ULN)
     4. ALT and AST < 5 × ULN
     5. Serum amylase and lipase ≤ 2 × ULN
     6. Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN
     7. Left ventricular ejection fraction of the heart is within the reference range
  8. Participants must meet the following criteria related to prior or current treatment:

     1. Patients on hydroxycarbamide for lowering cell counts: Discontinue hydroxycarbamide for at least 24 hours before initiating olverembatinib therapy
     2. Patients who have recurrence during cytotoxic therapy: Olverembatinib must be given at least 14 days after the last dose of chemotherapy with the following exceptions: Intrathecal (IT) chemotherapy and/or maintenance therapy, e.g., vincristine, purinethol, methotrexate, or glucocorticoids. For relapsed patients on maintenance therapy, 24-hour washout period is required.
     3. Hematopoietic stem cell transplantation (HSCT): Patients who relapse after HSCT are acceptable, provided that they do not have acute or chronic graft versus host disease (GVHD) or receive GVHD prophylaxis or treatment, and use the first dose of olverembatinib at least 90 days after transplantation.
     4. Biological and targeted drug products: At least a 7-day washout period is required for biological products prior to the first dose of olverembatinib. If a known adverse event (AE) occurs following the discontinuation of biological products, the period must be prolonged to cover the onset time of the known AE. The specific washout period can be comprehensively determined by the investigator.
     5. Monoclonal antibodies: There must be at least 3 half-lives from the use of monoclonal antibodies to the first dose of olverembatinib.
     6. Immunotherapy: Prior to the first dose of olverembatinib, there should be at least a 30-day washout period after completing any type of immunotherapies (e.g., tumor vaccine and chimeric antigen receptor T cell [CAR-T-cell]).
     7. Immunosuppressive therapy: Prior to the first dose of olverembatinib, there must be at least a 14-day washout period after completing immunosuppressive therapy (including the regimen after stem cell transplantation).
     8. Radiotherapy: No washout period is needed for the radiotherapy of any extramedullary site excluding the central nervous system (CNS); if subjects have received whole-body irradiation or craniospinal radiation or cranial radiation, the washout period must be more than 90 days.
     9. Anthracyclines: Prior to the first dose of olverembatinib, a cumulative dose of anthracyclines received by subjects must be less than 400 mg/m2 of adriamycin equivalent.
     10. Subjects who do not use concomitant medications that may have potential drug-drug interactions with olverembatinib. Or else, at least 5-day washout period is required.
     11. Subjects who never used olverembatinib.

Exclusion Criteria:

* The subject who meets any of the following criteria cannot be enrolled in this study:

  1. Any AEs (excluding alopecia and pigmentation) that are due to other anti-tumor therapies have not recovered to CTCAE v5.0 grade 0 - 1.
  2. Gastrointestinal dysfunction or gastrointestinal diseases that may significantly alter absorption of study drug.
  3. Uncontrollable or serious cardiovascular diseases.
  4. Subjects with symptomatic CNS disorder (e.g., convulsion caused by CNS disorder).
  5. Patients who have significant bleeding unrelated to Ph+ ALL.
  6. Patients who are known to have hypersensitivity to any component of the study drug.
  7. Patients with uncontrolled systemic infection, or there is laboratory or clinical evidence for infection with active human immunodeficiency virus, hepatitis B virus, hepatitis C virus, or SARS-CoV-2.
  8. Vaccination with attenuated live vaccines within 28 days prior to study treatment.
  9. Patients who have any conditions that, in the opinion of the investigator, would jeopardize the patient safety or interfere with the evaluation of safety and efficacy of the study drug.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 42 days
  DLT evaluation is defined as adverse events or laboratory abnormalities that occur within 6 weeks after investigational drug administration, are unrelated to external causes such as progressive disease, concomitant disease, and concomitant medications, including hematologic and non-hematologic adverse events (grade according to NCI CTCAE 5.0).
Objective Response Rate (ORR) | 132 days
  ORR is defined by Complete Remission (CR)+ CR with incomplete marrow recovery (CRi) + Partial Remission (PR).Response will be evaluated every period till complete treatment and three months after last dose.
Maximum plasma concentration (Cmax) | 42 days
  Maximum plasma concentration (Cmax) will be assessed on all participants of each dose group on the first day of olverembatinib monotherapy in period 1, and on the first and last days of olverembatinib in combination with APG-2575 in period 2 .
Area under the plasma concentration versus time curve (AUC) | 42 days
  Area under the plasma concentration versus time curve (AUC) will be assessed on all participantsof each dose group on the first day of olverembatinib monotherapy in period 1, and on the first and last days of olverembatinib in combination with APG-2575 in period 2 .
R2PD of Olverembatinib and APG-2575 | 42 days
  To confirm the recommended doses of olverembatinib and APG-2575 in children with Ph+ ALL

SECONDARY OUTCOMES:
Minimal Residual Disease (MRD) negative rate | 132 days
  To observe the proportion of subjects with MRD negative status in bone marrow.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Zhu, MD, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, CAMS & PUMC
Locations (4):
- China (4):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Department of Pediatrics, Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Department of Hematology/Oncology, Shanghai Jiaotong University School of Medicine Affiliated Shanghai Children's Medical Center, Shanghai

IPD SHARING:
Plan to Share IPD: No